CLINICAL TRIAL: NCT05313763
Title: The Effect of Kinesio Taping on Cervical Proprioception Sense, Pain, Disability and Quality of Life in Patients With Cervical Spondylosis
Brief Title: The Effect of Kinesio Taping With Cervical Spondylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Emre Ata, Assoc Prof, Associate Proffesor, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2194
Record Dates: First submitted 2022-03-23; First posted 2022-04-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Cervical Spondylosis
Keywords: Cervical Spondylosis; kinesio-tape; cervical proprioception
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional physical therapy group (Experimental): Conventional physical therapy is the first line of treatment in cervical spondylosis.
  Interventions: Other: conventional physical therapy
- Kinesio-tape Group (Active Comparator): Conventional rehabilitation program will be applied five days a week, 3 weeks, a total of 15 sessions. Kinesio-tape applications will be applied in 6 sessions during conventional physical therapy, twice a week at four-day intervals.
  Interventions: Other: conventional physical therapy; Other: Active Kinesiotaping
- Sham kinesio-tape Group (Sham Comparator): Conventional rehabilitation program will be applied five days a week, 3 weeks, a total of 15 sessions. Sham kinesio-tape applications will be applied twice a week at four-day intervals, 6 sessions during conventional physical therapy.
  Interventions: Other: conventional physical therapy; Other: Sham Kinesiotaping

INTERVENTIONS:
Other: conventional physical therapy — A hotpack will be applied to the neck area for 15 minutes in the prone position of the patients. Conventional type Tens with a frequency of 50 Hz and a pulse duration of <150 microseconds will be applied for 20 minutes, taking the painful area to the center. Ultrasound will be applied to the patients for 5 minutes with a dosage of 1-1.5 watts/cm2. Cervical joint range of motion exercises, stretching exercises for trapezius, scalenia, rhomboid, levator scapulae, pectoral and suboccipital muscles will be applied, then cervical isometric strengthening exercises and stabilization exercises will be carried out in a controlled manner. Conventional physical therapy will be applied by the same physiotherapist 5 days a week for 3 weeks.
Other: Active Kinesiotaping — For kinesio-tape application, a 20 cm long Y strip and a 15 cm long I strip tape will be prepared. The patient will flex his neck, and the application will be started from the midline of the upper thoracic vertebrae. Initially, 4-5 cm stretching will be applied, and the arms of the Y strip will be adhered to the cervical paravertebral muscles without stretching. I strip will be applied to the painful area with the area correction technique, with maximum stretching in the middle and without stretching the ends. The applications will be made by the same physiatrist with 7 years of clinical experience.
  Arms: Kinesio-tape Group
Other: Sham Kinesiotaping — For Sham kinesio-tape application, a 20 cm long Y strip and a 15 cm long I strip tape will be prepared. The patient will flex his neck, the application will be started from the midline of the upper thoracic vertebrae, and the Y and I bands will be applied without stretching. The applications will be made by the same physiatrist with 7 years of clinical experience.
  Arms: Sham kinesio-tape Group

SUMMARY:
The investigators aimed to evaluate the effect of kinesio tape application on the sense of proprioception in patients with cervical spondylosis.This research aims to determine the relationship between the sense of cervical proprioception and neck pain intensity, neck disability and quality of life, and to determine the relationship between cervical spinal MRI findings and cervical proprioception. Studies conducted to date are limited to the evaluation of patients who underwent kinesio tape for neck pain in terms of joint range of motion, pain, and disability. In a study examining the relationship between cervical kinesio-tape application and cervical proprioception sense; The patient group consists of the young population and the patient evaluation was made immediately after the end of the treatment. The aim of this study is to evaluate the relationship of kinesio tape applied to the elderly patient group with cervical spondylosis, where the cervical proprioception sense is more affected, with cervical proprioception sense in the mid-term and to examine its relationship with cervical spinal MRI phenotypes. The possible relationship between proprioceptive sensory deficit and joint degeneration is based on a combination of neuromuscular control dysfunction and periarticular degeneration. Thus, the investigators aimed to improve the proprioceptive sense, reduce pain and increase functionality in the elderly patient group with kinesio-tape in the study.

DETAILED DESCRIPTION:
Cervical spondylosis is the aging of the cervical spine as a result of degeneration of the intervertebral discs. In this process, shortening of the disc distance in the cervical spine, thickening of the ligaments, development of ligamentous and segmental instability, arthrosis and loss of lordosis in the facet joints are observed. Degenerative disc changes are often seen as bulging, protrusion, extrusion, and sequestration. Cervical discs are thicker anteriorly than posteriorly, resulting in normal lordosis. In the degenerative process, first of all, the height decreases in the anterior of the disc and loss of lordosis occurs. The process progresses with aging and causes axial neck pain and/or disc herniations due to degenerative changes, intraspinal canal and foraminal stenosis, secondary radiculopathy or myelopathy symptoms.

Although there is no complete consensus about the pathophysiological mechanism that causes cervical degenerative disc disease, several hypotheses have been developed. Although spondylosis is seen as a normal part of aging according to the current approach, certain occupations, repetitive movements and traumas can accelerate the process. Only a single factor has no chance to trigger the degenerative process. In other words, many factors of the normal aging process affect cervical spondylolysis. Although age-related degeneration is the primary cause, cervical disc injuries may affect this degenerative process in younger patients.

Degeneration in the cervical spine may only present with neck pain if there is no compression on the spinal cord or nerve root. This degeneration causes radicular pain in the occipital region, posterior neck, shoulder or arm due to inflammation due to extrinsic compression in the nerve root. Patients with cervical spondylosis usually present with complaints of pain, tingling, numbness, and weakness in the upper extremities, resulting in significant disability and functional limitations.

Proprioception is a sense of bodily movement position that includes a sense of joint position and a sense of movement (kinesthesia). Proprioceptive information reaches the central nervous system via the afferent pathway, which contributes to movement and postural neuromuscular control. The cervical muscles have an abundant muscle spindle density reflecting a rich proprioceptive system, which contributes to enhanced sensorimotor function and therefore plays an important role in maintaining effective motor control and static and dynamic postures.

Studies have shown that sense of cervical position is vital in maintaining joint stability under static and dynamic conditions, and impaired proprioception may predispose to the development of pain. Cervical proprioception is measured by joint position error in degrees. In cervical spondylosis, impaired cervical proprioception is the result of position sensitivity being affected primarily by impairment in the muscles, joints, or capsules and secondarily by changes in afferent proprioceptive adjustment and integration. Impaired position sense impairs both neuronal and muscular control of normal cervical joint function, resulting in unbalanced muscle strength and placing the joint at risk for trauma.

Conservative treatment of spondylosis includes transcutaneous electrical nerve stimulation (TENS), heat, traction, exercise, postural training, massage, kinesiotaping, and numerous manual therapy and mobilization techniques. Recent studies investigating treatment modalities for neck pain associated with cervical spondylosis have shown that combined treatments are more effective than exercise alone.

The kinesio-tape technique has been developed with the philosophy that positive results can be obtained with a taping method similar to the structural properties and flexibility of human skin, without limiting the joint movements of the kinesio tape. Latex-free kinesio-tape is composed of 100% cotton and elastic polymer fibers. Dr. According to Kase, muscle dysfunction is one of the leading problems originating from the musculoskeletal system. Dr. Kase argues that taping the muscle is more effective than immobilizing the joint circumference with tape. After injury or overuse, the elastic properties of the muscle deteriorate. For this reason, kinesiology tapes are designed to be similar to the elastic properties of the muscle, to be adhesive, to have a lifting effect on the skin to which kinesiology tapes are applied, and to allow air circulation between the skin and the external environment. The technique is based on 3 basic concepts. These are space, motion, and cooling. As painful and inflamed muscles swell due to edema, the area where muscles are located narrows. When kinesio-taping is applied, the skin and subcutaneous interstitial area are increased by lifting the skin, thus increasing circulation and movement. This reduces pain and improves performance. The neuromuscular system is retrained. Injuries are prevented, circulation is accelerated and tissue healing is ensured.

The idea that kinesiotaping can regulate proprioception by affecting cutaneous mechanoreceptors has been put forward by some researchers. Kinesiolo-tape affects mechanoreceptors sensitive to tension, loading, pressure and shear forces by changing the length of the skin and superficial fascia and the tension of the muscle fibers. This can lead to significant changes in muscle movement and tone. Slow pressure stimulation, particularly on connective tissue, alters the effect on mechanoreceptors and may affect gamma motor neuron firing and muscle tone regulation. Kinesiotape can be particularly effective in increasing proprioceptive ability only in the middle of the movement. In this range, ligament mechanoreceptors are inactive, whereas muscle receptors are active. Understanding joint movement and position can be effective in the development of proprioception by stimulating sensory afferent transmission. Cutaneous afferent stimuli interact with the motor cortex and thus affect the muscle excitability of the central nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Being over 50 and under 70
* Moderate to severe neck pain and limitation in neck movements according to the Visual Analogue Scale, which has been present for at least 3 months
* Presence of cervical degeneration radiologically
* being literate
* Giving consent by agreeing to participate in the study
* Having an MRI registered in the system in the last 1 (one) year

Exclusion Criteria:

* Being under 50 and over 70
* Neck pain that has been present for less than 3 months
* Patients with positive Spurling test and radiculopathy
* Patients with nerve root compression and stenosis in the evaluation with cervical MRI within the last 1 year
* History of neurological disease, history of neck trauma, cervical myelopathy, any inflammatory arthritis, tumor, infection involving the cervical spine, and vertebrobasilar artery insufficiency
* Cervical spinal surgery history
* Vestibular disorder
* vision problems
* cognitive impairment
* polyneuropathy
* B12 and vitamin D deficiency (Patients with abnormal values for B12 and vitamin D in the last three months through the hospital examination result system will not be included in the study)
* No known diagnosis of psychotic disorder
* Active skin infection, cellulitis, open wounds, presence of cancerous tissue, extreme obesity and allergy to adhesives containing polyacrylate
* not being literate
* Patients who received physical therapy, injection, manual therapy, kinesio-tape treatment from the neck region in the last 3 months.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
change in cervical proprioception after treatment | change in cervical proprioception will be evaluated 1 month after treatment
  It is measured by the cervical joint position error test. This test assesses whether the patient can return to the previous neutral position after maximum rotation of the head in the coronal and sagittal planes. A headlamp with a laser light source in the middle, an eye patch, a 40 cm diameter target with trigonometric segments, a metal and magnetic apparatus used to adjust the target according to its neutral position are used as equipment.The patient is seated in a chair with his eyes closed in a neutral position; The target is positioned at a distance of 90 cm. The target is a 40 cm diameter circle and contains five separate small circles to which the grading is applied. These small circles are called 1 degree, 2 degrees, 3 degrees, 4.5 degrees, and 6 degrees, which allows to evaluate the deviation. The target is adjusted according to the patient's height.

SECONDARY OUTCOMES:
cervical joint range of motion | Evaluations will be made before treatment, immediately after treatment, and 1 month after treatment.
  It is measured with a goniometer. While all movements of the neck are evaluated as active and passive, they are evaluated in terms of limitation and pain. Normal joint ranges of motion in the cervical region are: 80-90 degrees of flexion, 20-45 degrees of lateral flexion, 70 degrees of extension and 90 degrees of rotation.
Hand grip strength | Evaluations will be made before treatment, immediately after treatment, and 1 month after treatment.
  It will be evaluated with the Jamar hydraulic hand dynamometer.The purpose of this test is to test the maximum isometric contraction strength of the hand and forearm muscles. A hand grip dynamometer is required to perform the test (such as Jamar™, Camry™, Smedley™). Dynamometer Examples Grip strength should be evaluated while the patient is sitting in the chair. The elbows are kept close to the body and at 90° flexion. The wrist is in neutral. The person to be measured is asked to grasp the dynamometer and squeeze it as hard as he can. The test result is determined by calculating the average of the three measurements. Norm values for measurement: 47-40kg for men aged 20-69 (left hand 2 kg less) 30-24kg for women (1.5-2kg less for left hand),
Upper extremity functionality | Evaluations will be made before treatment, immediately after treatment, and 1 month after treatment.
  Upper extremity functionality to be measured by upper extremity functional index (UEFI).The Upper Extremity Functional Index was developed in 2001 to evaluate the functional disability of the upper extremity (50). The first version consists of 20 questions. There is also a version of the scale that was reduced to 15 questions after Rasch analysis (51.52). Aytar et al. In 2015, Turkish cultural adaptation, validity and reliability study was carried out. Scoring is calculated based on Likert scoring (0: extremely difficult/not able to do at all, 4: no difficulty). The scoring of the version consisting of 15 questions is between 0-100 points, and a high score indicates a high level of activity. This scale, which is specific to the region, is completed in about 5 minutes.
Neck pain | Evaluations will be made before treatment, immediately after treatment, and 1 month after treatment.
  Neck pain will be measured with the Visual Analog Scale (VAS).The Visual Analog Scale (VAS) is used to convert some values that cannot be measured numerically. Two end definitions of the parameter to be evaluated are written at the two ends of a 100 mm line, and the patient is asked to indicate where on this line their situation is appropriate by drawing a line or by placing a dot or pointing. For example, for pain, I have no pain at one end and very severe pain at the other end and the patient marks his/her current state on this line. The length of the distance from the point where there is no pain to the point marked by the patient indicates the patient's pain.
Neuropathic pain | Evaluations will be made before treatment, immediately after treatment, and 1 month after treatment.
  Neuropathic pain will be measured with the Douleur Neuropathique 4 Questions (DN4).Douleur neuropathique en 4 questions (DN4) asks 7 questions about symptoms and 3 questions about clinical management. The DN4 scoring is an easy tool and a total score of 4 or more out of 10 indicates neuropathic pain. With the same results, 7 sensory discriminators can be used as a self-report tool. DN4 has been shown to have 83% sensitivity and 90% specificity.
Neck disability | Evaluations will be made before treatment, immediately after treatment, and 1 month after treatment.
  Neck disability will be measured with the Neck Disability Index (NDI).This form consists of 10 questions. The intensity of pain in the neck, the difficulty in personal care, the ability to lift a load, the interaction of reading with neck pain, headaches, difficulty in doing work, driving, difficulty in sleeping and leisure activities are questioned. Each question scores between 0 and 5 points, and an increased score is associated with increased disability. If the volunteer does not drive, does not do leisure time activities and does not work in a job, these questions are calculated by subtracting them from the scoring. The neck disability rate of the patient is calculated by multiplying the score the volunteers get with the maximum score they can get, multiplied by 100. As this rate increases, it is accepted that the patient's neck-related disability increases.
SF-36 | Evaluations will be made before treatment, immediately after treatment, and 1 month after treatment.
  Quality of life will be measured with the 36-Item Short Form Survey (SF-36).The primary feature of the SF-36 is that it is a self-assessment scale. It is considered among the advantages of the scale that it can be filled in as little as five minutes, and that it can evaluate the positive as well as the negative aspects of the health status. The scale consists of 36 items and they provide the measurement of 8 dimensions; physical function (10 items), social function (2 items), role limitations due to physical functions (4 items), role limitations due to emotional problems (3 items), mental health (5 items), energy/vitality (4 items), pain (2 items) and general perception of health (5 items). The scale is evaluated considering the last 4 weeks. In order to create the acute form, a form evaluating the last 1 week was also applied.
Mood | Evaluations will be made before treatment, immediately after treatment, and 1 month after treatment.
  Mood will be measured with the Hospital Anxiety and Depression Scale (HAD).It is a self-assessment scale developed to determine the risk of anxiety and depression in patients with physical illness and those applying to primary health care services, and to measure its level and change in severity (Zigmond and Snaith 1983). It was translated into Turkish by Aydemir et al. and its validity and reliability study was conducted. It has anxiety and depression subscales. The internal consistency (Cronbach alpha) of the scale was 0.8525 for the anxiety subscale and 0.7784 for the depression subscale. The item-total score correlation coefficients ranged between 0.8161-0.8547 in the anxiety subscale and between 0.7374-0.7795 in the depression subscale. In two-half reliability, r=0.8532 for anxiety subscale and 0.8069 for depression subscale. It consists of 14 questions in total. The minimum score for the anxiety and depression subscales is 0, and the maximum score is 21.
Cervical spinal MRI | Evaluations will be made before treatment
  Cervical spinal MRI will be evaluated with Cervical Phenotype Index (CPI).It is an index that comprehensively evaluates degenerative cervical spine findings, and it has been found to be associated with patient-reported NDI and VAS, and is predictive of prognosis for operated patients. This index scores C2-T1 vertebrae on disc degeneration, disc space narrowing, disc displacement, Modic changes, end plate abnormalities (e.g. schmorl's nodules), high-density regions (HIZs), osteophytes.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Ata, Ass.Prof., Principal Investigator — Sultan II. Abdulhamidhan Training and Research Hospital
Locations (1):
- Sultan 2. Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Türkiye)